CLINICAL TRIAL: NCT00137527
Title: Prospective, Randomized Trial of Cerebral Oximetry Monitoring in Patients Undergoing Coronary Artery Bypass Surgery
Brief Title: Brain Oxygenation Monitoring in Patients Undergoing Coronary Artery Bypass Surgery
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Atlantic Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: B03-07-008
Record Dates: First submitted 2005-08-26; First posted 2005-08-30 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Neurological Manifestations
Keywords: Cardiac Surgery; Cardiopulmonary Bypass; Cerebral Oxygenation; Neurologic Dysfunction; Neurocognitive Dysfunction; Neurological manifestations; Memory loss; Delirium; Coronary Artery Bypass
MeSH Terms: conditions — Neurologic Manifestations; Cognition Disorders; Memory Disorders; Delirium

INTERVENTIONS:
Device: Optimizing hemodynamic and anesthetic parameters to improve cerebral perfusion

SUMMARY:
The purpose of this study is to determine whether intraoperative brain oxygenation monitoring in cardiac surgery patients is effective in reducing postoperative neurologic and neurocognitive dysfunction.

DETAILED DESCRIPTION:
This study represents a prospective, randomized assessment of the potential clinical and economic benefit to be derived from the continuous non-invasive monitoring of regional cerebral oxygen saturation (rSO2) during cardiac surgery employing cardiopulmonary bypass (CPB). Previous studies have shown that low rSO2 values obtained during surgery are highly associated with postoperative frontal lobe dysfunction, cognitive declines, disorientation, and other clinical indices of prolonged recovery. Low rSO2 values are thought to reflect the development of tissue hypoxia within susceptible regions of the cerebral cortex during the non-pulsatile perfusion of CPB. Rapid detection and correction of such episodes should help avoid regional hypoxia and its attendant postoperative sequelae. This study will assess neurologic, psychometric, and quality of life markers of brain dysfunction which could result from CPB. Each study patient will be assessed both pre- and postoperatively (pre-hospital discharge and at three months) for neurologic and neurocognitive dysfunction.

Comparison(s): Intervention versus control group. Patients assigned to the intervention rSO2-monitored group will be managed with conservative measures designed to maintain the rSO2 value at, or above, its preoperative value. Such measures include increases in pump flow, blood pressure, anesthetic dose, arterial oxygen tension, carbon dioxide tension, and hematocrit. Those patients in the control group will be managed according to current established practice. Although rSO2 is also recorded in this group, the monitor's readings are blinded.

ELIGIBILITY:
Inclusion Criteria:

* Primary coronary artery bypass surgery
* Ages 18-90
* Voluntary participation with signed informed consent

Exclusion Criteria:

* An unwillingness to participate in the study
* Inability to obtain informed consent
* Expressive or receptive aphasia
* Inability to correctly perform the neurocognitive tests preoperatively
* Inability to correctly perform the saccadic and anti-saccadic eye movement tests preoperatively
* Non-English speaking candidates
* Patients for whom it is known that follow-up will be improbable
* Previous cardiac surgery
* Concomitant procedures
* Pre-existing psychotic disorders
* Patients with active alcohol (ETOH) abuse requiring emergent surgery
* Patients scoring 2 or higher on the CAGE evaluation
* Mini-Mental State Exam preoperative score of 23 or less
* Severe visual or auditory disorders
* Parkinson's disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250
Dates: Start 2004-02; Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Cognitive function measured by neurocognitive tests administered in the preoperative, immediate postoperative, and three months postoperative periods

SECONDARY OUTCOMES:
Relationship of intraoperative risk data to postoperative cognitive function

CONTACTS AND LOCATIONS:
Overall Officials: James P Slater, MD, Principal Investigator — Morristown Memorial Hospital
Locations (1):
- Morristown Memorial Hospital, Morristown, New Jersey, United States

REFERENCES:
- [Background] Newman MF, Kirchner JL, Phillips-Bute B, Gaver V, Grocott H, Jones RH, Mark DB, Reves JG, Blumenthal JA; Neurological Outcome Research Group and the Cardiothoracic Anesthesiology Research Endeavors Investigators. Longitudinal assessment of neurocognitive function after coronary-artery bypass surgery. N Engl J Med. 2001 Feb 8;344(6):395-402. doi: 10.1056/NEJM200102083440601. PMID 11172175
- [Background] Selnes OA, Grega MA, Borowicz LM Jr, Royall RM, McKhann GM, Baumgartner WA. Cognitive changes with coronary artery disease: a prospective study of coronary artery bypass graft patients and nonsurgical controls. Ann Thorac Surg. 2003 May;75(5):1377-84; discussion 1384-6. doi: 10.1016/s0003-4975(03)00021-3. PMID 12735550
- [Background] Selnes OA, McKhann GM. Neurocognitive complications after coronary artery bypass surgery. Ann Neurol. 2005 May;57(5):615-21. doi: 10.1002/ana.20481. PMID 15852408